CLINICAL TRIAL: NCT01570166
Title: Percutaneous Radiofrequency Ablation Versus Repeat Hepatectomy for Recurrent Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, professor, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HCC16
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; RFA; HR
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA (Experimental): For RFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Interventions: Procedure: HR
- HR group (Experimental): HR was carried out under general anesthesia using a right subcostal incision with a midline extension.Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant, and the possibility of a negative resection margin. Anatomic resection, in the form of segmentectomy and/or subsegmentectomy as described by Makuuchi et al. (16) was the preferred surgical method of liver resection. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 min and 5 min, respectively; this technique was used repeatedly throughout the entire procedure. Hemostasis of the raw liver surface was done with suturing and application of fibrin glue.
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: HR — HR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant, and the possibility of a negative resection margin. Anatomic resection, in the form of segmentectomy and/or subsegmentectomy as described by Makuuchi et al. (16) was the preferred surgical method of liver resection. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 min and 5 min, respectively; this technique was used repeatedly throughout the entire procedure.
  Other Names: hepatic resection; surgical resection
  Arms: RFA
Procedure: RFA — For PRFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Other Names: percutenous ablation
  Arms: HR group

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world. Partial hepatectomy is still considered as the conventional therapy for HCC. Intrahepatic recurrence of HCC after partial hepatectomy is common and was reported to be more than 77% within 5 years after surgery. Repeat hepatectomy is an effective treatment for intrahepatic HCC recurrence, with a 5-year survival rate of 19.4-56%. This is comparable to the survival after initial hepatectomy for HCC. Unfortunately, repeat hepatectomy could be carried out only in a small proportion of patients with HCC recurrence (10.4-31%), either because of the poor functional liver reserve or because of widespread intrahepatic recurrence. In the past two decades, percutaneous radiofrequency ablation (PRFA) has emerged as a new treatment modality and has attracted great interest because of its effectiveness and safety for small HCC (≤ 5.0 cm). Studies using PRFA to treat recurrent HCC after partial hepatectomy reported a 3-year survival rate of 62-68%, which is comparable to those achieved by surgery. PRFA is particularly suitable to treat recurrent HCC after partial hepatectomy because these tumors are usually detected when they are small and PRFA causes the least deterioration of liver function in the patients. To the best of our knowledge, there has been no report published in the medical literature comparing the efficacy of repeat hepatectomy with PRFA for recurrent HCC. The aim of this retrospective study is to compare the outcome of repeat hepatectomy with PRFA for small recurrent HCC after partial hepatectomy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world. Partial hepatectomy is still considered as the conventional therapy for HCC. Intrahepatic recurrence of HCC after partial hepatectomy is common and was reported to be more than 77% within 5 years after surgery. Repeat hepatectomy is an effective treatment for intrahepaticHCC recurrence, with a 5-year survival rate of 19.4-56%. This is comparable to the survival after initial hepatectomy for HCC. Unfortunately, repeat hepatectomy could be carried out only in a small proportion of patients with HCC recurrence (10.4-31%), either because of the poor functional liver reserve or because of widespread intrahepatic recurrence. In the past two decades, percutaneous radiofrequency ablation (PRFA) has emerged as a new treatment modality and has attracted great interest because of its effectiveness and safety for small HCC (≤ 5.0 cm). Studies using PRFA to treat recurrent HCC after partial hepatectomy reported a 3-year survival rate of 62-68%, which is comparable to those achieved by surgery. PRFA is particularly suitable to treat recurrent HCC after partial hepatectomy because these tumors are usually detected when they are small and PRFA causes the least deterioration of liver function in the patients. To the best of our knowledge, there has been no report published in the medical literature comparing the efficacy of repeat hepatectomy with PRFA for recurrent HCC. The aim of this retrospective study is to compare the outcome of repeat hepatectomy with PRFA for small recurrent HCC after partial hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 75 years;
2. Distant recurrence of HCC after initial curative treatment (including initial RFA or hepatectomy);
3. no other treatment received except for the initial RFA or hepatectomy;
4. Single tumor less than 4cm in diameter;
5. lesions visible on ultrasound and with an acceptable and safe path between the lesion and the skin as shown on ultrasound;
6. no severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3;
7. Eastern Co-operative Oncology Group performance(ECOG) status 0 -

Exclusion Criteria:

1. the presence of vascular invasion or extrahepatic spread on imaging;
2. a Child-Pugh class C liver cirrhosis or evidence of hepatic decompensation including ascites, severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3), esophageal or gastric variceal bleeding or hepatic encephalopathy;
3. an American Society of Anesthesiologists (ASA) score ≥ 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5-year

SECONDARY OUTCOMES:
disease-free survival | 5-year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-set University, Guangzhou, Guangdong, China